CLINICAL TRIAL: NCT02470650
Title: Cost-effectiveness of Different Antiretroviral Treatment in Patients HIV Naive. Randomized Clinical, Not Masked, Trial Comparing DRVr3TC, ABC3TC (Kivexa) RPV, or EVG COBI FTC TDF (Stribild) for 48 Weeks
Brief Title: Cost-effectiveness of Different Antiretroviral Treatment in Patients HIV Naive
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Josep Mallolas, Principal Investigator, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cost-Effect-Clinic; 2014-004820-24 (EudraCT Number)
Record Dates: First submitted 2015-05-29; First posted 2015-06-12 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Patient Compliance; Antiretroviral Therapy Intolerance
Keywords: comparative effectiveness
MeSH Terms: conditions — Patient Compliance | interventions — elvitegravir; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Darunavir; abacavir, lamivudine drug combination; Ritonavir; Lamivudine; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- elvitegravir/cobicistat/emtricitabine/tenofovir (Experimental): EVG / COBI / FTC / TDF (Stribild®) 150 elvitegravir, 150 cobicistat, 200 emtricitabine, 245 tenofovir disoproxil. 1 recovered tablet once a day (on a day)
  Interventions: Drug: elvitegravir/cobicistat/emtricitabine/tenofovir
- darunavir+ritonavir+lamivudine (Active Comparator): Darunavir 800 mg (Prezista®) 1 recovered tablet once a day Ritonavir 100 mg(Norvir® ) 1recovered tablet once a day lamivudine300 mg (Epivir®) 1 recovered tablet once a day
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Lamivudine
- abacavir/lamivudine+rilpivirine (Active Comparator): Abacavir 600 mg +lamivudine 300mg (Kivexa®) 1tablet once a day rilpivirine (Edurant®) 1 recovered tablet 25 mg. once a day
  Interventions: Drug: abacavir/lamivudine; Drug: rilpivirine

INTERVENTIONS:
Drug: elvitegravir/cobicistat/emtricitabine/tenofovir — 1 recovered tablet once Per day ● Specify total dose (number and unit): 150 mg de elvitegravir, 150 mg cobicistat, 200 mg emtricitabine , 245 mg tenofovir disoprox milligram(s)
  Other Names: Stribild
  Arms: elvitegravir/cobicistat/emtricitabine/tenofovir
Drug: Darunavir — Darunavir 800 mg (Prezista®) 1 recovered tablet 800 mg once a day
  Other Names: prezista
  Arms: darunavir+ritonavir+lamivudine
Drug: abacavir/lamivudine — Abacavir 600 mg /lamivudine 300 mg recovered tablet once a day
  Other Names: Kivexa
  Arms: abacavir/lamivudine+rilpivirine
Drug: Ritonavir — Ritonavir 100 mg recovered tablet once a day
  Other Names: Norvir
  Arms: darunavir+ritonavir+lamivudine
Drug: Lamivudine — lamivudine 300mg (Epivir) 1 recovered tablet
  Other Names: Epivir
  Arms: darunavir+ritonavir+lamivudine
Drug: rilpivirine — rilpivirine (Edurant®) 1 recovered tablet 25 mg. once a day
  Other Names: Edurant
  Arms: abacavir/lamivudine+rilpivirine

SUMMARY:
The main objective of this study is to know the efficiency (costeffectiveness) at 48 weeks of initiation of antiretroviral treatment. three strategies of treatment.

DETAILED DESCRIPTION:
Secondary objectives:

* patients with virologic response ratio at 48 weeks (less than 50 plasma viral load)
* Change in the number of CD4 cells at 48 weeks
* Change in body composition and mineral density bone (body and lumbar) measurement with DEXA (bone mineral density scan) at 48 weeks
* Change in markers of renal function (creatinine clearance, glomerular filtration rate - eGFR - estimated rate) and renal tubular function at 48 weeks
* Rate of mortality and clinical progression at 48 weeks
* general tolerability and safety: adverse events (AA) and serious AA description

ELIGIBILITY:
Inclusion Criteria:

* 1-negative pregnancy test in women of childbearing age
* 2- stable HIV-1 infection clinically and not take antiretroviral therapy
* 3- viral load HIV <100,000 copies
* 4- CD4 cells >100 cels/mm3
* 5- Glomerular filtration >70mlmin
* 6- have a negative HLA B5701
* 7-.patients should have given informed written consent
* 8- in the opinion of the investigator, be able to follow the design of the Protocol visits

Exclusion Criteria:

* 1-. Patients who had virologic failure with any antiretroviral therapy
* 2- evidence of prior mutations of the study drugs
* 3- use of any anti-retroviral treatment in the 6 months prior to the entry of the study
* 4- contraindication to the drugs study
* 5- any condition that does not allow to ensure the correct compliance to the study
* 6- uncontrolled previous psychiatric illness
* 7- Current or active addiction or alcoholism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
efficiency (cost-effectiveness) | 48 weeks of initiation antiretroviral treatment
  Antiretroviral treatment effectiveness defined by the number of patients with <37 copies/ml viral load at the 48 weeks and the treatment cost defined by the sum of cost ogfthe antiretroviral treatment and all its consequences (adverse effects, changes of pattern study antiretroviral resistance in case of being necessary, days of sick leave by the patient and hospital admission days) that occur in the 48 weeks. The price of the antiretroviral treatment will be defined by Spanish official price.

SECONDARY OUTCOMES:
Change in the number of CD4 cells | 48 weeks
  Change in the number of CD4 cells at 48 weeks
number of patients with virologic response ratio copies mL plasma viral load) | 48 weeks
  less than 37 copies/mL in plasma viral load
Change in body composition and mineral density bone lumbar) measurement with DEXA | 48 weeks
  Measurement baseline and at 48 weeks. DEXA Scan (Dual X-ray Absorptiometry) to Measure Bone Health
Change in markers of renal function filtration rate - eGFR - estimated rate) and renal tubular function | 48 weeks
  Defined by creatinine clearance, glomerular filtration rate - eGFR - and renal tubular function at week 48 filtration rate - eGFR - estimated rate) and renal tubular function at 48 weeks

OTHER OUTCOMES:
Rate of mortality and clinical progression | 48 weeks
  Defined by diagnostic AIDS diseases or death

CONTACTS AND LOCATIONS:
Overall Officials: Mallolas, Principal Investigator — Hospital Clínic

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT02470650/Prot_SAP_000.pdf